CLINICAL TRIAL: NCT00218478
Title: Cue Reactivity Model for Assessing Pharmacologic Intervention in Treatment of Cannabis Use Disorders (Study 1)
Brief Title: Evaluating Responses to Drug-Related Cues Versus Neutral Cues to Understand the Effects of Marijuana Craving - 1
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Leslie Lundahl, Principal Investigator, Wayne State University
Other Study IDs: NIDA-19236-1; R21DA019236-01 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Marijuana Abuse
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Cue Desensitization — During the study session, both groups will be shown a nature video and will be asked to handle and smell various items; these will act as the neutral, non marijuana-related cues. Next, the participants will watch a video of individuals smoking marijuana and will be asked to handle and smell marijuana-related items; these will act as the marijuana-related cues.

SUMMARY:
The majority of past research on marijuana treatment has specifically targeted the alleviation of withdrawal symptoms. Minimal focus has been placed on how altering craving effects may play a role in treating marijuana addiction. The purpose of this study is to compare the effects of marijuana-related cues versus non marijuana-related cues in individuals both addicted and not addicted to marijuana. In turn, this may help establish a better understanding of the effects of marijuana cravings and may lead to improved treatments for marijuana dependence.

DETAILED DESCRIPTION:
Marijuana is the most commonly used illegal drug in the United States; more than 2 million Americans either abuse or are dependent on the drug. The development of a medication to reduce marijuana use and prevent drug relapse by lessening withdrawal symptoms has been a primary focus of research. However, there has been little emphasis on evaluating the efficacy of a treatment that specifically reduces marijuana cravings. This study will evaluate the subjective and physiological responses to marijuana-related cues versus non marijuana-related cues in order to better understand the effects of marijuana cravings.

Participants will be divided into two groups. Group 1 will consist of 20 individuals diagnosed with marijuana dependence; Group 2 will consist of individuals matched by age range, gender and race to Group 1, and who are healthy volunteers and do not use marijuana or who report limited marijuana exposure. Participants in Group 1 will spend one night at the Psychiatric and Addiction Research Center at Detroit Receiving Hospital to control for alcohol and drug use for 12 hours preceding the next day's 2-hour study session. Participants in Group 2 are not required to spend the night, but are tested for drugs and alcohol prior to the session. During the study session, both groups will be shown a nature video and will be asked to handle and smell various items; these will act as the neutral, non marijuana-related cues. Next, the participants will watch a video of individuals smoking marijuana and will be asked to handle and smell marijuana-related items; these will act as the marijuana-related cues. Heart rate and skin temperature will be monitored continuously throughout the cue sessions with the use of electrodes and a skin thermometer. Prior to and after the cue sessions, blood pressure will be measured and questionnaires will be administered to assess drug cravings as well as related mood states. Prior to leaving the laboratory, the participants' vital signs will be evaluated to ensure that any cue-related physiological changes have returned to normal. Participants will have the option of talking to a clinician experienced in dealing with drug cravings following the end of the study session.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnosis criteria for marijuana dependence. Participants enrolled in the control group should not meet DSM-IV diagnosis criteria for any Axis I disorder, and should not use marijuana or have had limited marijuana exposure.
* Reads and writes English
* If female, willing to use adequate contraception throughout the study

Exclusion criteria:

* Meets DSM-IV diagnosis criteria for a psychiatric illness
* History of a psychotic disorder
* Seeking treatment for marijuana dependence
* Neurologic disease, including structural brain abnormalities (e.g., neoplasms), stroke, seizures, infectious disease, head trauma resulting in unconsciousness, or evidence of neurologic illness resulting from HIV/AIDS
* Cardiovascular disease, including edema, chest pain or palpitations after exertion or drug use, myocardial infarction (heart attack), systolic blood pressure greater than 160 mmHg or less than 95 mmHg, or diastolic blood pressure greater than 95 mmHg
* Pulmonary disease, including apnea, cor pulmonale, tuberculosis, dyspnea, orthopnea, or tachypnea
* Systemic disease, including endocrinopathies, kidney or liver failure, hypothyroidism, adrenocortical insufficiency, or an autoimmune disease involving the central nervous system
* Currently dependent on any drug other than marijuana or nicotine
* Cognitively impaired
* Pregnant or breastfeeding

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Marijuana dependent volunteers
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2004-09; Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie H. Lundahl, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Lundahl LH, Greenwald MK. Magnitude and duration of cue-induced craving for marijuana in volunteers with cannabis use disorder. Drug Alcohol Depend. 2016 Sep 1;166:143-9. doi: 10.1016/j.drugalcdep.2016.07.004. Epub 2016 Jul 18. PMID 27436749